CLINICAL TRIAL: NCT04991935
Title: A Phase 3, Multicenter, Multinational, Open-Label Extension Study to Evaluate the Long-Term Safety of CC-93538 in Adult and Adolescent Subjects With Eosinophilic Esophagitis
Brief Title: Safety Study of CC-93538 in Adult and Adolescent Participants With Eosinophilic Esophagitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-93538-EE-002; 2020-004335-24 (EudraCT Number)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; CC-93538; RPC4046; Adult; Adolescent; Gastrointestinal Diseases; Esophagitis; Gastroenteritis; Eosinophils; Eosinophilia; Esophageal Diseases; Allergic Diseases; Antibody, Monoclonal; Hypersensitivity; Immunologic factors; Physiological Effects of Drugs; Cendakimab
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastrointestinal Diseases; Esophagitis; Gastroenteritis; Eosinophilia; Esophageal Diseases; Hypersensitivity | interventions — cendakimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-93538 (Experimental): Participants are administered CC-93538 dose subcutaneously once weekly
  Interventions: Drug: CC-93538

INTERVENTIONS:
Drug: CC-93538 — CC-93538
  Other Names: BMS-986355; cendakimab

SUMMARY:
This study is an open-label, uncontrolled study design to evaluate the long-term safety and tolerability of treatment with CC-93538. The study will enroll participants who participated in the CC-93538-EE-001 or CC-93538-DDI-001 studies.

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in prior clinical study CC-93538-EE-001 and either:

  1. Subject experienced a severe EoE flare requiring endoscopic intervention and/or concomitant rescue therapy during the Induction Phase and has completed Week 24 of the Induction Phase; OR
  2. Subject completed the Induction Phase and does not qualify for entry to the Maintenance Phase for reasons other than a severe EoE flare; OR
  3. Subject experienced a severe EoE flare requiring endoscopic intervention and/or concomitant rescue therapy during the Maintenance Phase and completed Week 48 of the Maintenance Phase; OR
  4. Subject completed Week 48 of the Maintenance Phase
* OR Subject must have participated in Study CC-93538-DDI-001 and completed assessments through the end of treatment visit
* Demonstrated ≥ 80% and ≤ 120% overall compliance with required investigational product dosing during the prior studies.
* Did not permanently discontinue investigational product in the prior studies and/or did not experience any clinically significant adverse events related to Investigational Product that would preclude further dosing in the opinion of the Investigator.
* Females of childbearing potential must have a negative pregnancy test prior to the first dose of open-label CC-93538 and agree to practice a highly effective method of contraception (as defined in the prior study) until 5 months after the last dose of open-label CC-93538.

Exclusion Criteria:

* Clinical or endoscopic evidence of other diseases or conditions that may affect or confound the histologic, endoscopic, or clinical symptom evaluation for this study.
* Active Helicobacter pylori infection or esophageal varices.
* Evidence of immunosuppression, or of having received systemic immunosuppressive or immunomodulating drugs within 5 drug half-lives prior to open-label extension study (OLE) Day 1. Use of these agents is prohibited during the study.
* Treatment with oral or sublingual immunotherapy within 6 months of OLE Day 1. Use of these agents is prohibited during the study.
* Received an investigational product, other than that administered in the CC-93538-EE-001 or CC-93538-DDI-001 studies, within 5 half-lives prior to OLE Day 1 (includes investigational product received during an interventional trial for COVID-19). Those vaccinated with an investigational COVID-19 vaccine during the CC-93538-EE-001 or CC-93538-DDI-001 studies are not eligible to participate, unless allowed following a discussion with the Clinical Trial Physician.
* Received a live attenuated vaccine within one month prior to OLE Day 1; or anticipates the need for a live attenuated vaccine at any time throughout the course of this study.
* Any disease that would affect the conduct of the protocol or interpretation of the study results, or would put a patient at risk by participating in the study (e.g. colitis, celiac disease, Mendelian disorder associated with EoE, severe uncontrolled asthma, infection causing eosinophilia, hypereosinophilic syndrome, or cardiovascular condition, or neurologic or psychiatric illness that could compromise the participant's ability to accurately document symptoms of EoE; newly diagnosed malignancy, lymphoproliferative disease, or clinically significant laboratory abnormality).
* Active parasitic/helminthic infection or a suspected parasitic/helminthic infections or chronic infection (viral hepatitis, tuberculosis, or HIV)
* Has had idiopathic anaphylaxis or major immunologic reaction to an immunoglobulin-G containing agent; or any known hypersensitivity to any ingredient in CC-93538.
* Females who are pregnant or lactating.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | For a minimum of 28 months
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

SECONDARY OUTCOMES:
Immunogenicity of CC-93538 assessed through the incidence of anti-drug antibodies | For a minimum of 28 months
  This includes neutralizing antibodies when warranted.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (167):
- United States (81):
  - Local Institution - 144, Birmingham, Alabama
  - Local Institution - 082, Phoenix, Arizona
  - Local Institution - 147, Phoenix, Arizona
  - Local Institution - 041, Scottsdale, Arizona
  - Local Institution - 029, Tucson, Arizona
  - Local Institution - 165, North Little Rock, Arkansas
  - Local Institution - 075, Lancaster, California
  - Local Institution - 047, Los Angeles, California
  - Local Institution - 160, San Diego, California
  - Local Institution - 068, Aurora, Colorado
  - Local Institution - 067, Colorado Springs, Colorado
  - Local Institution - 128, Wheat Ridge, Colorado
  - Local Institution - 101, Bristol, Connecticut
  - Local Institution - 076, Farmington, Connecticut
  - Local Institution - 156, Hamden, Connecticut
  - Local Institution - 099, Clearwater, Florida
  - Local Institution - 036, Inverness, Florida
  - Local Institution - 042, Jacksonville, Florida
  - Local Institution - 138, Miami, Florida
  - Local Institution - 146, Orlando, Florida
  - Local Institution - 169, Pinellas Park, Florida
  - Local Institution - 168, Plantation, Florida
  - Local Institution - 037, Port Orange, Florida
  - Local Institution - 171, Atlanta, Georgia
  - Local Institution - 054, Atlanta, Georgia
  - Local Institution - 117, Macon, Georgia
  - Local Institution - 024, Idaho Falls, Idaho
  - Local Institution - 039, Chicago, Illinois
  - Local Institution - 167, Gurnee, Illinois
  - Local Institution - 127, Clive, Iowa
  - Local Institution - 094, Iowa City, Iowa
  - Local Institution - 035, Kansas City, Kansas
  - Local Institution - 046, Florence, Kentucky
  - Local Institution - 003, Baton Rouge, Louisiana
  - Local Institution - 020, Metairie, Louisiana
  - Local Institution - 044, Metairie, Louisiana
  - Local Institution - 164, Columbia, Maryland
  - Local Institution - 070, Glen Burnie, Maryland
  - Local Institution - 012, Hagerstown, Maryland
  - Local Institution - 053, Boston, Massachusetts
  - Local Institution - 083, South Dartmouth, Massachusetts
  - Local Institution - 009, Worcester, Massachusetts
  - Local Institution - 014, Wyoming, Michigan
  - Local Institution - 115, Plymouth, Minnesota
  - Local Institution - 049, Rochester, Minnesota
  - Local Institution - 007, Kansas City, Missouri
  - Local Institution - 032, St Louis, Missouri
  - Local Institution - 038, Omaha, Nebraska
  - Local Institution - 015, Lebanon, New Hampshire
  - Local Institution - 139, Albuquerque, New Mexico
  - Local Institution - 028, Great Neck, New York
  - Local Institution - 051, New York, New York
  - Local Institution - 116, Syracuse, New York
  - Local Institution - 142, Syracuse, New York
  - Local Institution - 016, Chapel Hill, North Carolina
  - Local Institution - 106, Durham, North Carolina
  - Local Institution - 131, Greensboro, North Carolina
  - Local Institution - 130, Beavercreek, Ohio
  - Local Institution - 006, Cincinnati, Ohio
  - Local Institution - 001, Cincinnati, Ohio
  - Local Institution - 052, Cincinnati, Ohio
  - Local Institution - 059, Columbus, Ohio
  - Local Institution - 166, Oklahoma City, Oklahoma
  - Local Institution - 120, Hershey, Pennsylvania
  - Local Institution - 025, Philadelphia, Pennsylvania
  - Local Institution - 155, Pottsville, Pennsylvania
  - Local Institution - 143, Anderson, South Carolina
  - Local Institution - 057, Greenville, South Carolina
  - Local Institution - 114, Chattanooga, Tennessee
  - Local Institution - 095, Nashville, Tennessee
  - Local Institution - 105, Cedar Park, Texas
  - Local Institution - 148, Dallas, Texas
  - Local Institution - 112, Houston, Texas
  - Local Institution - 008, San Antonio, Texas
  - Local Institution - 077, Southlake, Texas
  - Local Institution - 104, Tyler, Texas
  - Local Institution - 125, Ogden, Utah
  - Local Institution - 013, Lynchburg, Virginia
  - Local Institution - 064, Richmond, Virginia
  - Local Institution - 137, Spokane, Washington
  - Local Institution - 023, Vancouver, Washington
- Argentina (2):
  - Local Institution - 695, Mar del Plata
  - Local Institution - 696, Quilmes
- Australia (14):
  - Local Institution - 548, Concord, New South Wales
  - Local Institution - 554, Liverpool, New South Wales
  - Local Institution - 540, Westmead, New South Wales
  - Local Institution - 546, Maroorchydore, Queensland
  - Local Institution - 550, South Brisbane, Queensland
  - Local Institution - 542, Woolloongabba, Queensland
  - Local Institution - 552, Adelaide, South Australia
  - Local Institution - 545, Elizabeth Vale, South Australia
  - Local Institution - 553, Clayton, Victoria
  - Local Institution - 543, Footscray, Victoria
  - Local Institution - 539, Melbourne, Victoria
  - Local Institution - 549, Murdoch, Western Australia
  - Local Institution - 538, Fitzroy
  - Local Institution - 547, Western Australia
- Austria (3):
  - Local Institution - 437, Burgenland
  - Local Institution - 434, Graz
  - Local Institution - 436, Linz
- Belgium (4):
  - Local Institution - 515, Brussels
  - Local Institution - 516, Kortrijk
  - Local Institution - 514, Leuven
  - Local Institution - 512, West-Vlaanderen
- Canada (7):
  - Local Institution - 201, Calgary, Alberta
  - Local Institution - 208, Edmonton, Alberta
  - Local Institution - 205, Edmonton, Alberta
  - Local Institution - 203, Vancouver, British Columbia
  - Local Institution - 206, Victoria, British Columbia
  - Local Institution - 207, Ottawa, Ontario
  - Local Institution - 200, Vaughan, Ontario
- Germany (5):
  - Local Institution - 330, Bayern
  - Local Institution - 332, Brandenburg
  - Local Institution - 339, Frankfurt am Main
  - Local Institution - 338, Leipzig
  - Local Institution - 337, München
- Israel (6):
  - Local Institution - 278, Tel Aviv, Tel Aviv
  - Local Institution - 281, Haifa
  - Local Institution - 283, Holon
  - Local Institution - 280, Jerusalem
  - Local Institution - 282, Jerusalem
  - Local Institution - 279, Ẕerifin
- Italy (5):
  - Local Institution - 257, Genova
  - Local Institution - 254, Milan
  - Local Institution - 255, Padua
  - Local Institution - 252, Pisa
  - Local Institution - 253, Rome
- Japan (12):
  - Local Institution - 600, Nishinomiya, Hyōgo
  - Local Institution - 595, Bunkyo-ku, Tokyo
  - Local Institution - 599, Setagaya-ku, Tokyo
  - Local Institution - 593, Akita
  - Local Institution - 606, Isehara City, Kanagawa
  - Local Institution - 597, Kobe
  - Local Institution - 598, Maebashi
  - Local Institution - 607, Nagoya
  - Local Institution - 603, Okayama
  - Local Institution - 602, Shinjuku-Ku
  - Local Institution - 605, Tokyo
  - Local Institution - 590, Yamagata
- Poland (10):
  - Local Institution - 385, Bydgoszcz
  - Local Institution - 389, Częstochowa
  - Local Institution - 390, Gdansk
  - Local Institution - 388, Katowice
  - Local Institution - 392, Lódz
  - Local Institution - 387, Warsaw
  - Local Institution - 393, Warsaw
  - Local Institution - 383, Warsaw
  - Local Institution - 391, Wroclaw
  - Local Institution - 384, Wroclaw
- Portugal (4):
  - Local Institution - 307, Lisbon
  - Local Institution - 305, Lisbon
  - Local Institution - 306, Porto
  - Local Institution - 308, Porto
- Spain (6):
  - Local Institution - 408, Barcelona
  - Local Institution - 410, Córdoba
  - Local Institution - 409, Madrid
  - Local Institution - 413, Madrid
  - Local Institution - 411, Marbella
  - Local Institution - 412, Seville
- Local Institution - 357, Lausanne, Switzerland
- United Kingdom (7):
  - Local Institution - 228, Belfast Northern Ireland
  - Local Institution - 231, Birmingham
  - Local Institution - 234, Cardiff
  - Local Institution - 235, Chorley
  - Local Institution - 233, Hexam
  - Local Institution - 236, Liverpool
  - Local Institution - 237, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com